CLINICAL TRIAL: NCT07368738
Title: Intravenous Acetaminophen and Ketorolac for Pain Management During Extracorporeal Shockwave Lithotripsy: A Randomized Controlled Trial
Brief Title: Intravenous Acetaminophen and Ketorolac for Pain Management During Extracorporeal Shockwave Lithotripsy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Horizon Health Network (Other)
Responsible Party: Principal Investigator, Sufyan Faridi, Principal Investigator, Horizon Health Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6191
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Extracorporeal Shockwave Lithotripsy
Keywords: acetaminophen; ketorolac; extracorporeal shockwave lithotripsy; intravenous; pain
MeSH Terms: conditions — Pain | interventions — Midazolam; Fentanyl; Acetaminophen; Ketorolac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid (Active Comparator)
  Interventions: Drug: IV midazolam; Drug: IV fentanyl
- Non-Opioid (Experimental)
  Interventions: Drug: IV midazolam; Drug: IV acetaminophen; Drug: IV ketorolac

INTERVENTIONS:
Drug: IV midazolam — 1-2 mg
Drug: IV fentanyl — 25-300 mcg
  Arms: Opioid
Drug: IV acetaminophen — 1 g
  Arms: Non-Opioid
Drug: IV ketorolac — 30 mg
  Arms: Non-Opioid

SUMMARY:
The goal of this clinical trial is to learn if a non-opioid pain medicine regimen works as well as or better than a standard opioid-based regimen to manage pain during extracorporeal shockwave lithotripsy (ESWL) in adults.

The main questions it aims to answer are: Does the non-opioid regimen lead to similar or better pain control during the procedure? Does the non-opioid regimen lead to similar or better procedure tolerability and side effect profile?

The non-opioid regimen will use intravenous (IV) midazolam plus IV acetaminophen and IV ketorolac, and the standard opioid-based regimen will use IV midazolam plus IV fentanyl.

Participants will be randomly assigned to receive one of the two medication regimens during ESWL, and asked to rate their pain before the procedure and 30 minutes after the procedure.

DETAILED DESCRIPTION:
Extracorporeal shockwave lithotripsy (ESWL) is a common outpatient treatment for renal and ureteric stones, but the shockwaves can be painful and often require intra-procedure sedation and analgesia to improve comfort and allow delivery of an adequate number of shockwaves at therapeutic energy settings. Opioid-based regimens are widely used for ESWL because they are familiar, titratable, and effective; however, peri-procedural opioid exposure is increasingly scrutinized in the context of Canada's opioid crisis.

This study is a prospective randomized controlled trial in adults undergoing ESWL at St. Joseph's Hospital in Saint John, New Brunswick. The trial compares an opioid-sparing, multimodal regimen (intravenous midazolam, acetaminophen, and ketorolac) with a standard opioid-based regimen (intravenous midazolam and fentanyl). The primary objective is to evaluate the effectiveness of the non-opioid multimodal regimen on procedural pain compared with the standard opioid-based regimen. Secondary objectives include comparing shockwave tolerability and the adverse effect profile between regimens.

Participants are randomly allocated to a regimen and remain blinded to which regimen they receive. Sedation/analgesia is administered intravenously according to the assigned pathway, with midazolam titrated to achieve moderate sedation and analgesia provided via fentanyl (opioid arm) or a multimodal combination of ketorolac and acetaminophen (non-opioid arm).

Pain is measured using a 0-10 numeric rating scale (NRS). The NRS is administered before ESWL and 30 minutes after ESWL. Procedure tolerability is assessed using proxy measures recorded during ESWL (total shockwaves delivered and highest energy level achieved). Adverse medication effects recorded include hypotension, oxygen desaturations, and nausea/vomiting.

The overarching goal is to determine whether an opioid-sparing ESWL pathway can provide equal or superior pain control while maintaining comparable procedural tolerability and safety, supporting routine adoption of non-opioid multimodal analgesia when feasible.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Undergoing ESWL
* Able to provide informed consent

Exclusion Criteria:

* Prior ESWL treatment in the past six months
* Narcotic use in the last 48 hours
* Allergy to midazolam, fentanyl, acetaminophen, or ketorolac
* Chronic kidney disease
* Solitary kidney
* Active peptic ulcer disease
* Concurrent anticoagulant prescription
* Liver disease
* Elevated liver function tests
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pain as Assessed by the NRS | Before the procedure, and 30 minutes after the procedure
  The numeric rating scale (NRS) will be used to quantify pain. Scores range from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Procedure Tolerability as Assessed by Total Number of Shockwaves Delivered and Highest Energy Level Achieved | During the procedure
Rate of Adverse Medication Effects | During the procedure
  Hypotension, oxygen desaturations, nausea/vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Whelan, MD, FRCSC, Principal Investigator — Department of Urology - Horizon Health Network
Locations (1):
- St. Joseph's Hospital, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No